CLINICAL TRIAL: NCT04861675
Title: Assessment of Changes in Oral Health-related Quality of Life , Oral Hygiene Status and Body Growth in Egyptian Children With Special Health Care Needs Following Dental Treatment Under General Anaesthesia
Brief Title: Assessment of Changes in Oral Health-related Quality of Life , Oral Hygiene Status and Body Growth in CSHCN Following Dental Treatment Under General Anaesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahy Abdel Raouf Aly Kamar, Principal Investigator, Cairo University
Other Study IDs: 14422019465983
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Quality of Life; General Anesthesia; Children With Special Health Care Needs; Body Mass Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective follow up cohort study: Assessment of Changes in Oral Health-related Quality of Life , Oral Hygiene status and Body Growth in Egyptian Children with Special Health Care Needs following Dental Treatment under General Anaesthesia
  Interventions: Procedure: Full mouth rehabilitation under general anaesethia

INTERVENTIONS:
Procedure: Full mouth rehabilitation under general anaesethia — Assessment of change in oral health related quality of life , body growth status and oral hygiene status for children with special health care needs after full mouth rehabilitation under general anesethia,

SUMMARY:
evaluation of the impact of dental treatment under GA on oral health-related quality of life (OHRQoL) in children with SHCN with severe dental caries with Assessment in change in oral health status and the impact on children's weight (Wt), height (Ht), Body Mass Index (BMI).

DETAILED DESCRIPTION:
The study consisted of clinical dental examinations performed at the time of DGA and at the six-month recall, along with OHRQoL questionnaires and data drawn from the patients' files.

1. OHRQoL will be assessed with the early childhood oral health impact scale (ECHOIS) that is composed of items which assess the effect of oral health condition on different aspects of life of the patient .
2. Children with Mental special health care needs will be recruited from G.A unit in department of pediatric dentistry , faculty of oral and dental medicine cairo university.
3. Data will be collected for each of the study participants included age, gender ,Medical (type of disability and history of disability) , dental histories and clinical findings were correlated accordingly together with determining the type of disability, anthropometric measures (HT, WT,BMI) that will be measured at baseline and after 3 to 6 months from dental treatment under general anesthesia.
4. The parent or the care giver will be taken as a surrogate measure that will self-complete (ECOHIS) Before and after treatment with follow up after 3 & 6 months to assess and evaluate children's OHRQoL and anthropometric measures update.
5. Each GA session included a comprehensive clinical dental examination and full dental rehabilitation. The Silness-Loe plaque index (PI) was used to assess oral hygiene status. That was measured in the four levels of distal facial, mesial-facial, facial, and lingual of first molars, first premolar and central in each quadrant using mirror and probe.
6. The plaque index was obtained by adding the figures of the four above-mentioned areas of each teeth and dividing it by 4 before recording it in the examination form
7. Parents/ caregiver will be asked to consider the last 6 months when responding the questions After ttt , Examine effect of oral rehabilitation under GA and its effect on improving quality of life ( pain , eating problems, sleeping problems ,growth parameters as (Wt, Ht, BMI) and any postoperative complications as postoperative pain and pharynx discomfort or fever

ELIGIBILITY:
Inclusion Criteria:

* Intellectual disabled children with carious teeth

Exclusion Criteria:

* Healthy children
* children with physical special needs.
* Refusal of participation.
* Participation in any other concurrent clinical trials.
* Presence of any serious medical condition or transmissible diseases such as hepatitis , AIDS or malignancies.
* Children whose parents refuse to sign the consent or have no phone no. to enable post-operative contact.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Mental special health care needs undergoing oral rehabilitation under general anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in oral health related quality of life. | 6 months
  Early childhood oral health impact scale , A total score of ECOHIS ranging from 0 to 52 was calculated as a simple sum of the responses. Higher scores representing a greater oral health impact and/or poorer OHRQoL.

SECONDARY OUTCOMES:
Oral hygiene status | 6 months
  Plaquei ndex (Löe and Silness, 1963)

OTHER OUTCOMES:
Body mass index | 6 months
  weight and height will be combined to report BMI in kg/m^2

IPD SHARING:
Plan to Share IPD: No